CLINICAL TRIAL: NCT03820102
Title: Impact of Metabolic Changes and Vitamin D Status on Virological Response in Patients With Hepatitis C Viral Infection Treated by Direct Acting Antiviral Drugs
Brief Title: Impact of Metabolic Changes and Vitamin D Status on Virological Response in Patients With HCV Infection Treated by DAAs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Hassan Abdelgawad, Gastroenterologest and hepatologest, doctor in Assiut Police Hospital, Assiut University
Other Study IDs: IR,VitD in HCV
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: HCV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vit D deficiency: Chronic HCV patients with vitamin D deficiency Sustained virological response after treatment
- Normal Vit D: Chronic HCV patients with normal vitamin D level Sustained virological response after treatment

SUMMARY:
1. Study Changes in lipid profile and the impact of Insulin resistance on virological response in patients with Hepatitis C viral infection treated by Direct Acting Antiviral agents
2. The assessment of serum vitamin D levels in HCV infected patients and predictive value of pre-treatment serum vitamin D level for achieving sustained virological response at 12 weeks post-treatment

DETAILED DESCRIPTION:
Patients and methods:

This cross-sectional study will include 100patients of chronic HCV infection who attend El Raghy Assiut university Hospital, either inpatients or outpatients. Chronic HCV infection will be diagnosed based on detectable HCV RNA with anti-HCV Ab in patient with clinical and/or ultrasonographic criteria of chronic liver disease.

Patients will receive treatment to HCV by DAAs and follow up for 12 weeks to confirm sustained virological response

Method:

Patients presenting in this study will be subjected to the following:

1. Full history and clinical evaluation.
2. Body weight (kg) and height (m).
3. BMI will calculate as weight divided by squared height (kg/m2).
4. Waist circumference will measured at a level midway between the lowest rib and the iliac crest, and the hip circumference at the level of the great trochanters, with the legs close together.
5. Blood pressure (mmHg) was measured twice in the upper arm after a 10-min period of rest and taken an average.

Laboratory investigations will include:

* Complete blood count (CBC)
* Liver function test
* HCV Ab and HCV RNA by PCR
* HBs Ag
* Alpha fetoprotein
* Lipid profile
* Serum urea and creatinine
* Fasting blood sugar (FBG)and Serum fasting insulin level
* Insulin resistance determined via Homeostasis Model Assessment (HOMA-IR) IR = fasting insulin (µu/ml) × fasting glucose (mmol/L) ----------------------------------------------------------------- 22.5 An index value of ˃ 2. 5 was defined as IR (Huang et al., 2011)
* Vitamin D level:

Vitamin D deficiency wasdefined as a 25 (OH)-vitamin D serum level < 20 ng/mL, vitaminD insufficiency as 25 (OH)-vitamin D levels of 20 - 29.9ng/mL, and normal vitamin D levels ≥ 30 ng/mL (Holick MF et al.,2011)

* Abdominal Ultrasound
* Electrocardiogram (ECG)

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV will receive DAAs for treatment

Exclusion Criteria:

1. Decompensated liver cirrhosis, hepatocellular carcinoma, history of liver transplant
2. Co-existing liver disease (hepatitis B virus, autoimmune hepatitis, human immunodeficiency virus)
3. Extra-hepatic malignancy except after two years of disease free interval.
4. Patients with diabetes mellitus.
5. Patients with Chronic kidney disease.
6. Pregnancy or in ability to use effective contraception.
7. Patients with history of using lipid lowering therapy
8. relapser or failure of previous HCV treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Full history and clinical evaluation.
  2. Body weight and height
  3. BMI will calculate as weight divided by squared height (kg/m2)
  4. Waist circumference
  5. Blood pressure (mmHg)
  Laboratory investigations will include:
  * Complete blood count (CBC)
  * Liver function test
  * HCV Ab and HCV RNA by PCR
  * HBs Ag
  * Alpha fetoprotein
  * Lipid profile
  * Serum urea and creatinine
  * Fasting blood sugar and Serum fasting insulin level
  * Insulin resistance determined via Homeostasis Model Assessment (HOMA-IR) IR = fasting insulin (µu/ml) × fasting glucose (mmol/L)
  22.5 An index value of ˃ 2. 5 was defined as IR (Huang et al., 2011)
  * Vitamin D level:
  * Abdominal Ultrasound
  * Electrocardiogram
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
SVR12 | 12 week after treatment
  sustained virological response 12 week after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Laila Abd Elbaky, profesor, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Janovy J Jr. Problems in the comparative physiology of some trypanosomatid flagellates. Acta Trop. 1977 Jun;34(2):177-84. PMID 19960
- [Result] Selhub J, Rosenberg IH. Demonstration of high-affinity folate binding activity associated with the brush border membranes of rat kidney. Proc Natl Acad Sci U S A. 1978 Jul;75(7):3090-3. doi: 10.1073/pnas.75.7.3090. PMID 28521
- [Result] Ramachandran N, Colman RF. Evidence for a critical glutamyl and an aspartyl residue in the function of pig heart diphosphopyridine nucleotide dependent isocitrate dehydrogenase. Biochemistry. 1977 Apr 19;16(8):1564-73. doi: 10.1021/bi00627a006. PMID 15585